CLINICAL TRIAL: NCT01687751
Title: Dexmedetomidine Compared to Midazolam for Symptom Control in Advanced Cancer Patients: A Pilot Randomized Controlled Trial (RCT)
Brief Title: Pilot Study Comparing Treatment With Dexmedetomidine to Midazolam for Symptom Control in Advanced Cancer Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study design determined to be not likely feasible
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FHREB 2012-057
Record Dates: First submitted 2012-08-29; First posted 2012-09-19 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2013-01

CONDITIONS: Pain Intractable; Delirium; Dyspnea; Nausea
Keywords: feasibility studies; conscious sedation/; dexmedetomidine/; midazolam/; infusions, subcutaneous/; palliative care/; terminal care/; terminally ill/; neoplasms/; treatment outcome; Precedex; "end of life"; Dying; Advanced cancer; mood/delirium/delirious
MeSH Terms: conditions — Pain, Intractable; Delirium; Dyspnea; Nausea; Neoplasms; Death | interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine 0.2 to 1.1 mcg/kg/hr by continuous subcutaneous infusion for up to 10 days
  Interventions: Drug: Dexmedetomidine
- Midazolam (Active Comparator): Midazolam 10 to 100 mcg/kg/hr by continuous subcutaneous infusion for up to 10 days
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Dexmedetomidine — Study drugs will be administered by continuous subcutaneous infusion using a weight based protocol at a rate between 1.0 to 5.5 mL/hr.
  * The study drug will be started at a rate of 1.0 mL/hr.
  * The infusion rate is incremented by 0.5 ml/hr every 30 minutes until acceptable symptom control, bradycardia (heart rate < 40) or hypotension (systolic blood pressure < 80) prevent further increase or maximum infusion rate of 5.5 ml/hr, whichever comes first. Achievement of acceptable symptom control will be defined, for purposes of this trial, as a consensus between reports from patient, family care giver and attending registered nurse
  Other Names: Precedex; DIN 02339366
  Arms: Dexmedetomidine
Drug: Midazolam — Study drugs will be administered by continuous subcutaneous infusion using a weight based protocol at a rate between 1.0 to 5.5 mL/hr.
  * The study drug will be started at a rate of 1.0 mL/hr.
  * The infusion rate is incremented by 0.5 ml/hr every 30 minutes until acceptable symptom control, bradycardia (heart rate < 40) or hypotension (systolic blood pressure < 80) prevent further increase or maximum infusion rate of 5.5 ml/hr, whichever comes first. Achievement of acceptable symptom control will be defined, for purposes of this trial, as a consensus between reports from patient, family care giver and attending registered nurse
  Other Names: DIN 02240286
  Arms: Midazolam

SUMMARY:
Cancer patients with very difficult to control symptoms at the Abbotsford (AC) and Fraser Valley (FVC) Cancer Centers are referred and admitted to the Tertiary Palliative Care Units at the Abbotsford Regional Hospital and Cancer Center(ARHCC). For symptom management, patients are sometimes given midazolam continuously through a needle placed underneath the skin. While effective in symptom management, midazolam can be sedating, leaving patients unable to interact with loved ones in their last days.

This study is a pilot project. Before proceeding to a full-scale study, a "pilot study" or "feasibility study" is often carried out first to test the design of a study, the likelihood of successful recruitment or the acceptability of the intervention to potential subjects. The basic idea is to find out whether it will be practical to proceed to a larger study that will include more subjects. This type of study involves only a small number of subjects and therefore the results can only be used as a guide for further larger studies.

The investigators also will determine whether palliative care cancer patients taking a medication called dexmedetomidine would have improved rousability (more easily and fully awakened) and symptom control (pain, shortness of breath, nausea or confusion) compared with those taking standard of care which is receiving the medication midazolam. The use of dexmedetomidine in other clinical situations (in the Operating Room or Intensive Care Unit where the patient can still respond to the doctor) has been shown to be effective in symptom control and to provide a better degree of rousability to patients but has not been well studied in the palliative care environment.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND

Advanced cancer patients nearing the end of life suffer from pain, anxiety and other symptoms that can be very difficult to control. The current practice within Fraser Health Authority is to admit these patients to one of three tertiary palliative care units (TPCUs) for pain and symptom management. Once admitted, if pain and symptom relieving measures are insufficient, patients are given a continuous subcutaneous infusion (CSCI) of the drug midazolam for symptom management. While effective, sedation with midazolam often leaves patients unable to eat or drink or interact with their environment.

Dexmedetomidine is a unique and promising agent for managing intractable symptoms in palliative patients at the end of life . In addition to providing proportional sedation for symptom control, compared to midazolam, dexmedetomidine has the additional attributes of providing improved management of pain, dyspnea and delirium. Of special interest to patients who would like to continue to be involved in decision making and to be able to communicate with loved ones at the end of life is the quality of rousability possible when dexmedetomidine is used for sedation instead of midazolam. These features have been well studied in the ICU and anaesthesia literature but not in the palliative care environment.

PURPOSE AND JUSTIFICATION

Currently, standard care for patients with difficult or intractable symptoms for patients admitted to the tertiary palliative care units in Fraser Health is the administration of midazolam by CSCI as recommended in the evidence based Fraser Health Authority (FHA) Hospice Palliative Care Program Symptom Guideline "Refractory Symptoms and Palliative Sedation Therapy Guideline". The same guideline states that among the criteria for implementation of palliative sedation therapy is that "in all but the most unusual circumstances, death is anticipated within hours to days". However, many other patients with difficult or intractable symptoms have a natural course of their illness that is longer than 'hours to days'. These patients would benefit from a degree of sedation that is proportional to the severity of their symptoms. Therefore, particularly in these circumstances, an option other than deep palliative sedation with midazolam is necessary where the patient would very often like to be aware of those around them and still not be confused or in pain.

Despite many studies among ICU and anaesthesia patients, only two reports with four patients have evaluated use of dexmedetomidine in the palliative care environment. The first case was a 45 year old man with cervical paraganglioma, palliative performance scale (PPS) 10% with uncontrolled pain, insomnia, anxiety and severe psychological distress. Combined with morphine, a continuous intravenous infusion (CIVI) of dexmedetomidine provided relief of pain and anxiety within 30 minutes. The patient was sleeping without sign of pain, but prompt communication with his sister was possible. The infusion continued 24 hrs with good physical and psychological symptom control. The second case was 54 year old woman with breast cancer, PPS 20%, delirium and hypercalcemia. Treatment also included CIVI morphine, haloperidol 10 mg/day. Dexmedetomidine CIVI for 48 hr infusion improved agitation and the patient was able to transfer out of the bed, sit in a chair and communicate when necessary. When intravenous access was lost, the patient was sedated with midazolam CSCI 5 mg/hr and died 72 hours hours later. The third case was a 40 year old woman with advanced cervical cancer, PPS 10%, renal failure, hypercalcemia, intractable agitated delirium and pain with movement. Treatment included CSCI morphine, hydration and haloperidol 8 mg/day. Dexmedetomidine infusion temporarily improved delirium for 5 hours, but not pain with movement. When restlessness returned, dexmedetomidine was changed to midazolam 12 mg/hr for the 4 days until the patient died. The fourth case was a 46 year old woman with intractable back and left abdominopelvic pain radiating into her left leg. She was diagnosed with adenocarcinoma of unknown primary with a progressively expanding left retroperitoneal mass involving the psoas muscle and adjacent vertebral bodies. After the titration phase of dexmedetomidine, pain decreased to 6/10 as measured by a numerical pain scale which was considered tolerable by the patient. There was no significant sedation. By the third day, the pain increased to 9/10. As it was the patient's wish to go home, instead of up titrating the dexmedetomidine, a continuous epidural was started with bupivicaine and clonidine.

Current ongoing studies of dexmedetomidine use in the palliative care environment is limited to a Phase II study of dexmedetomidine in treating symptoms of distress in advanced cancer patients. The objective of this nine patient cohort study at Duke University Medical Center is to assess the effectiveness of 3 separate doses of dexmedetomidine (0.7, 1.5, 2.5 mg/kg/hr by continuous intravenous infusion) as add-on treatment for intractable pain, agitation and or delirium in terminally ill cancer patients in their last week of life until death. Overall, there is limited evidence in the literature to guide practice of using dexmedetomidine in the palliative care environment.

Given this gap in knowledge, the investigators propose to conduct a pilot randomized controlled trial (RCT) of dexmedetomidine CSCI compared to midazolam CSCI in advanced cancer patients in the palliative care setting.

The subcutaneous route is chosen for this pilot study as the preferred route of drug delivery as this conforms to the current standard of care according the FHA Hospice Palliative Care symptom guideline "Refractory Symptoms and Palliative Sedation Therapy Guideline": "Where feasible, the use of midazolam by CSCI is preferred to permit responsive titration. In general, subcutaneous administration is preferred to intravenous administration because of the practical advantage of subcutaneous infusion and the greater risk of apnea when bolus injections are administered intravenously". "The subcutaneous route is the most commonly used parenteral route in palliative care", "Drugs given via the subcutaneous route tend to have a high bioavailability (generally near 100 %)" "Subcutaneous infusion provides blood levels comparable to those from intravenous administration", "Perfusion of subcutaneous tissue is similar to that of muscle, but rate of absorption is slower."

Dexmedetomidine has been successfully administered by CSCI in the pediatric population, but so far has not been used by CSCI in palliative care patients. Neither midazolam or dexmedetomidine are currently approved for use by the subcutaneous route, but Health Canada approval will be obtained for the subcutaneous (SC) route for both dexmedetomidine and midazolam before starting the study to provide for use of the preferred subcutaneous route (over intravenous) in the palliative care environment. The goal of this trial is to assess the feasibility and methodological issues before enrolling subjects in a larger, multi-centre RCT to assess the effectiveness of dexmedetomidine in controlling pain, dyspnea, nausea and/or delirium compared to midazolam. Altogether, findings from this research program (pilot RCT and multi-centre RCT) will provide critical information for both clinicians and health policy makers on the use of dexmedetomidine in patients with advanced cancer with difficult to control or intractable symptoms.

RESEARCH QUESTION:

The overall goal of the investigators is to answer the following question: Does dexmedetomidine enhance control of pain, dyspnea, nausea and/or delirium, but with improved rousability, compared to midazolam in patients with advanced cancer? However, for the purposes of this pilot study, the investigators will address the following question: What is the feasibility of a multicentre RCT comparing dexmedetomidine with midazolam in enhancing control of pain, dyspnea, nausea and/or delirium in advanced cancer patients?

RESEARCH OBJECTIVE(S):

The objectives of this pilot study are:

* To identify facilitators and barriers to recruiting and consenting palliative care advanced cancer patients
* To assess site irritation when administering dexmedetomidine by continuous subcutaneous infusion as an alternate route to continuous intravenous infusion in advanced cancer patients
* To assess feasibility of collecting study measures
* To assess utility of a new study measurement of acceptable improvement of symptoms as assessed by patient, family, and staff

Other objectives of interest are:

* To compare arousability of palliative care advanced cancer patients when symptoms are controlled with dexmedetomidine as compared to midazolam
* To compare pain, dyspnea, nausea, delirium symptoms of palliative care advanced cancer patients sedated with dexmedetomidine as compared to midazolam

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 19 years of age
* Advanced cancer patient admitted to the Abbotsford Tertiary Palliative Care Unit
* Difficult to control or intractable symptom (REF 38, page 3)
* Midazolam CSCI would normally be considered for symptom management
* Informed consent is able to be provided in the English language
* Goals of care include do not resuscitate (DNR)
* For intractable symptoms, patient would prefer proportional sedation rather than no sedation or total sedation.

Exclusion Criteria:

* Second or third degree heart block (without pacemaker)
* Uncompensated congestive heart failure
* Heart rate less than 50 beats per minute
* Mean arterial blood pressure (MAP) < 60
* Weight below 35 kg. or above 85 kg.
* Prior use within the preceding 14 days of high dose benzodiazepines equivalent to the use of 30 mg or more of midazolam or 6 mg or more of lorazepam per 24 hours.
* Currently enrolled in any other research study involving drugs or devices

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects needed to recruit for a multicenter double blind randomized controlled phase III trial comparing dexmedetomidine to midazolam for symptom control in advanced cancer patients | one year
  Sample size determination for significant improvement in:
  * Pain
  * Dyspnea
  * Nausea
  * Delirium
  * Rousability

SECONDARY OUTCOMES:
Change in pain (0 to 10 numerical scale) | Up to 10 days
  Pain will be evaluated using the Edmonton Symptom Assessment Scale (ESASr)
Change in dyspnea (0 to 10 numerical scale) | Up to 10 days
  Dyspnea will be evaluated using the Edmonton Symptom Assessment Scale (ESASr)
Change in nausea (0 to 10 numerical scale) | Up to 10 days
  Nausea will be evaluated using the Edmonton Symptom Assessment Scale (ESASr)
Change in delirium (16 item clinician rated scale) | Up to 10 days
  Delirium will be assessed using the Delirium Rating Scale-Revised-98 (DRS-R-98)
Rousability (10 point scale) | Up to 10 days
  Rousability will be measured using the Richmond Agitation and Sedation Scale (RASS)
Acceptable symptom control (yes/no) | Up to 10 days
  Acceptable symptom control of the difficult to control or intractable symptoms of pain, dyspnea, nausea or delirium will be assessed by a two part question addressed to each of subject, family member and assigned palliative care nurse. Subjective responses will be collected from each as binary variables (0/1) with two positive responses indicating acceptable symptom control overall.

OTHER OUTCOMES:
Time to enroll 20 subjects | One year
  This information will be used to determine accrual rate. The accrual rate and the primary outcome measure of number needed to recruit will be used to determine the number of sites required for a multi-center double blind randomized controlled Phase III trial comparing dexmedetomidine to midazolam for symptom control in advanced cancer patients.
Cost determination for developing a budget for a large multi-center trial | One year

CONTACTS AND LOCATIONS:
Overall Officials: Neil K Hilliard, MD, Principal Investigator — 1. BC Cancer Agency 2. Fraser Health Authority; Stuart Brown, MD, Principal Investigator — Fraser Health Authority
Locations (1):
- Abbotsford Regional Hospital and Cancer Center, Abbotsford, British Columbia, Canada

REFERENCES:
- [Background] Abernethy AP. Pain and palliative care pharmacotherapy literature summaries and analyses. J Pain Palliat Care Pharmacother. 2008;22(2):145-51. doi: 10.1080/15360280801992140. PMID 19042839
- [Background] Anger KE, Szumita PM, Baroletti SA, Labreche MJ, Fanikos J. Evaluation of dexmedetomidine versus propofol-based sedation therapy in mechanically ventilated cardiac surgery patients at a tertiary academic medical center. Crit Pathw Cardiol. 2010 Dec;9(4):221-6. doi: 10.1097/HPC.0b013e3181f4ec4a. PMID 21119342
- [Background] Arain SR, Ruehlow RM, Uhrich TD, Ebert TJ. The efficacy of dexmedetomidine versus morphine for postoperative analgesia after major inpatient surgery. Anesth Analg. 2004 Jan;98(1):153-158. doi: 10.1213/01.ANE.0000093225.39866.75. PMID 14693611
- [Background] Brinkkemper T, van Norel AM, Szadek KM, Loer SA, Zuurmond WW, Perez RS. The use of observational scales to monitor symptom control and depth of sedation in patients requiring palliative sedation: a systematic review. Palliat Med. 2013 Jan;27(1):54-67. doi: 10.1177/0269216311425421. Epub 2011 Nov 1. PMID 22045725
- [Background] Caraceni A, Simonetti F. Palliating delirium in patients with cancer. Lancet Oncol. 2009 Feb;10(2):164-72. doi: 10.1016/S1470-2045(09)70018-X. PMID 19185834
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Cheung CW, Ying CL, Chiu WK, Wong GT, Ng KF, Irwin MG. A comparison of dexmedetomidine and midazolam for sedation in third molar surgery. Anaesthesia. 2007 Nov;62(11):1132-8. doi: 10.1111/j.1365-2044.2007.05230.x. PMID 17924894
- [Background] Chrysostomou C, Schmitt CG. Dexmedetomidine: sedation, analgesia and beyond. Expert Opin Drug Metab Toxicol. 2008 May;4(5):619-27. doi: 10.1517/17425255.4.5.619. PMID 18484919
- [Background] Clark, S., & Ezra, M. Use of dexmedetomidine as a sedative and analgesic agent in critically ill adult patients. Journal of the Intensive Care Society, 12(3), 244-245, 2011.
- [Background] Coull JT, Jones ME, Egan TD, Frith CD, Maze M. Attentional effects of noradrenaline vary with arousal level: selective activation of thalamic pulvinar in humans. Neuroimage. 2004 May;22(1):315-22. doi: 10.1016/j.neuroimage.2003.12.022. PMID 15110021
- [Background] Coyne PJ, Wozencraft CP, Roberts SB, Bobb B, Smith TJ. Dexmedetomidine: exploring its potential role and dosing guideline for its use in intractable pain in the palliative care setting. J Pain Palliat Care Pharmacother. 2010 Dec;24(4):384-6. doi: 10.3109/15360288.2010.518227. PMID 21133747
- [Background] Dere K, Sucullu I, Budak ET, Yeyen S, Filiz AI, Ozkan S, Dagli G. A comparison of dexmedetomidine versus midazolam for sedation, pain and hemodynamic control, during colonoscopy under conscious sedation. Eur J Anaesthesiol. 2010 Jul;27(7):648-52. doi: 10.1097/EJA.0b013e3283347bfe. PMID 20531094
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Gerlach AT, Murphy CV, Dasta JF. An updated focused review of dexmedetomidine in adults. Ann Pharmacother. 2009 Dec;43(12):2064-74. doi: 10.1345/aph.1M310. PMID 19934395
- [Background] Guinter JR, Kristeller JL. Prolonged infusions of dexmedetomidine in critically ill patients. Am J Health Syst Pharm. 2010 Aug;67(15):1246-53. doi: 10.2146/ajhp090300. PMID 20651314
- [Background] Jackson KC 3rd, Wohlt P, Fine PG. Dexmedetomidine: a novel analgesic with palliative medicine potential. J Pain Palliat Care Pharmacother. 2006;20(2):23-7. PMID 16702133
- [Background] Jones GM, Murphy CV, Gerlach AT, Goodman EM, Pell LJ. High-dose dexmedetomidine for sedation in the intensive care unit: an evaluation of clinical efficacy and safety. Ann Pharmacother. 2011 Jun;45(6):740-7. doi: 10.1345/aph.1P726. Epub 2011 Jun 10. PMID 21666095
- [Background] Kehl KA. Treatment of terminal restlessness: a review of the evidence. J Pain Palliat Care Pharmacother. 2004;18(1):5-30. PMID 15148006
- [Background] Kent CD, Kaufman BS, Lowy J. Dexmedetomidine facilitates the withdrawal of ventilatory support in palliative care. Anesthesiology. 2005 Aug;103(2):439-41. doi: 10.1097/00000542-200508000-00028. No abstract available. PMID 16052127
- [Background] Kunisawa T. Dexmedetomidine hydrochloride as a long-term sedative. Ther Clin Risk Manag. 2011;7:291-9. doi: 10.2147/TCRM.S14581. Epub 2011 Jul 11. PMID 21845052
- [Background] Lum, K. L., & Sanders, H. G. A comparison of midazolam and flunitrazepam in end-of-life care. Progress in Palliative Care, 19(1), 1-6, 2011.
- [Background] Maldonado JR, Wysong A, van der Starre PJ, Block T, Miller C, Reitz BA. Dexmedetomidine and the reduction of postoperative delirium after cardiac surgery. Psychosomatics. 2009 May-Jun;50(3):206-17. doi: 10.1176/appi.psy.50.3.206. PMID 19567759
- [Background] Maze M, Angst MS. Dexmedetomidine and opioid interactions: defining the role of dexmedetomidine for intensive care unit sedation. Anesthesiology. 2004 Nov;101(5):1059-61. doi: 10.1097/00000542-200411000-00002. No abstract available. PMID 15505438
- [Background] Mercadante S, Intravaia G, Villari P, Ferrera P, David F, Casuccio A. Controlled sedation for refractory symptoms in dying patients. J Pain Symptom Manage. 2009 May;37(5):771-9. doi: 10.1016/j.jpainsymman.2008.04.020. Epub 2008 Nov 28. PMID 19041216
- [Background] Muttu S, Liu EH, Ang SB, Chew PT, Lee TL, Ti LK. Comparison of dexmedetomidine and midazolam sedation for cataract surgery under topical anesthesia. J Cataract Refract Surg. 2005 Sep;31(9):1845-6. doi: 10.1016/j.jcrs.2005.09.019. No abstract available. PMID 16246802
- [Background] Prommer E. Review article: dexmedetomidine: does it have potential in palliative medicine? Am J Hosp Palliat Care. 2011 Jun;28(4):276-83. doi: 10.1177/1049909110389804. Epub 2010 Dec 3. PMID 21131636
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Roberts SB, Wozencraft CP, Coyne PJ, Smith TJ. Dexmedetomidine as an adjuvant analgesic for intractable cancer pain. J Palliat Med. 2011 Mar;14(3):371-3. doi: 10.1089/jpm.2010.0235. Epub 2011 Jan 17. PMID 21241196
- [Background] Ruokonen E, Parviainen I, Jakob SM, Nunes S, Kaukonen M, Shepherd ST, Sarapohja T, Bratty JR, Takala J; "Dexmedetomidine for Continuous Sedation" Investigators. Dexmedetomidine versus propofol/midazolam for long-term sedation during mechanical ventilation. Intensive Care Med. 2009 Feb;35(2):282-90. doi: 10.1007/s00134-008-1296-0. Epub 2008 Sep 16. PMID 18795253
- [Background] Shehabi, Y., Botha, J. A., Ernest, D., Freebairn, R. C., Reade, M., Roberts, B. L., et al. Clinical application, the use of dexmedetomidine in intensive care sedation. Critical Care and Shock, 13(2), 40-50, 2010.
- [Background] Soares LG, Naylor C, Martins MA, Peixoto G. Dexmedetomidine: a new option for intractable distress in the dying. J Pain Symptom Manage. 2002 Jul;24(1):6-8. doi: 10.1016/s0885-3924(02)00423-2. No abstract available. PMID 12183087
- [Background] Tan JA, Ho KM. Use of dexmedetomidine as a sedative and analgesic agent in critically ill adult patients: a meta-analysis. Intensive Care Med. 2010 Jun;36(6):926-39. doi: 10.1007/s00134-010-1877-6. Epub 2010 Apr 8. PMID 20376429
- [Background] Tobias JD. Subcutaneous dexmedetomidine infusions to treat or prevent drug withdrawal in infants and children. J Opioid Manag. 2008 Jul-Aug;4(4):187-91. doi: 10.5055/jom.2008.0024. PMID 18837201
- [Background] Trzepacz PT, Mittal D, Torres R, Kanary K, Norton J, Jimerson N. Validation of the Delirium Rating Scale-revised-98: comparison with the delirium rating scale and the cognitive test for delirium. J Neuropsychiatry Clin Neurosci. 2001 Spring;13(2):229-42. doi: 10.1176/jnp.13.2.229. PMID 11449030
- [Background] Ustun Y, Gunduz M, Erdogan O, Benlidayi ME. Dexmedetomidine versus midazolam in outpatient third molar surgery. J Oral Maxillofac Surg. 2006 Sep;64(9):1353-8. doi: 10.1016/j.joms.2006.05.020. PMID 16916668
- [Background] Wallace S, Mecklenburg B, Hanling S. Profound reduction in sedation and analgesic requirements using extended dexmedetomidine infusions in a patient with an open abdomen. Mil Med. 2009 Nov;174(11):1228-30. doi: 10.7205/milmed-d-00-6009. PMID 19960834
- [Background] Fraser Health Authority (FHA) Hospice Palliative Care Program Symptom Guideline "Refractory Symptoms and Palliative Sedation Therapy Guideline", May 9, 2011. Retrieved from http://www.fraserhealth.ca/media/RefractorySymptomsandPalliativeSedationTherapyRevised_Sept%2009.pdf )
- [Background] Flanagan E, Gentry J. He's taking how much Dilaudid! Dexmedetomidine: a novel approach to refractory symptom management. Presentation of the American Academy of Hospice and Palliative Medicine & Hospice and Palliative Nurses Association Conference 2011 Feb 16-19; Vancouver, British Columbia
- [Background] Doyle, D. et al, Oxford Textbook of Palliative Medicine, Third Edition 2004, p. 219.
- [Background] Storey P, Knight C. Assessment and Treatment of Pain in the Terminally Ill. UNIPAC Three, Hospice/Palliative Care Training for Physicians, A Self-Study Program, American Academy of Hospice and Palliative Medicine, Second Edition, Mary Ann Liebert, Inc., 2003, p. 62.